CLINICAL TRIAL: NCT00379977
Title: Open, Primary Vaccination Study to Assess Safety and Reactogenicity of GSK Biologicals' DTPa/Hib Vaccine When Administered to Healthy Chinese Infants at 3, 4 and 5 Months of Age.
Brief Title: Study to Assess the Safety & Reactogenicity of GSK Biologicals' DTPa/Hib Vaccine When Given at 3, 4 and 5 Months of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 106345
Record Dates: First submitted 2006-09-22; First posted 2006-09-25 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Tetanus; Haemophilus Influenzae Type b; Acellular Pertussis; Diphtheria
MeSH Terms: conditions — Tetanus; Haemophilus Infections; Diphtheria | interventions — Tetanus Toxoid; HibTITER protein, Haemophilus influenzae

INTERVENTIONS:
Biological: diphtheria, tetanus, pertussis & Hib vaccine
  Other Names: diphtheria; tetanus; pertussis & Hib vaccine

SUMMARY:
This study will evaluate the safety and reactogenicity of GSK Biologicals' Diphtheria Tetanus acellular Pertussis/Haemophilus influenzae type b vaccine given to Chinese infants at 3, 4 and 5 months of age.

ELIGIBILITY:
Inclusion Criteria:

* A male or female between, and including, 90 and 120 days of age at the time of the first vaccination Written informed consent obtained from the parent or guardian of the subject

Exclusion Criteria:

* subjects with known exposure to diphtheria, tetanus, pertussis and/or Haemophilus influenzae disease can not participate, subjects who have received previous vaccination against diphtheria, tetanus, acellular pertussis and/or Haemophilus influenzae type b (Hib) diseases can not participate.

Ages: 90 Days to 120 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30
Dates: Start 2006-09; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited symptoms during the 4 days following vaccination, unsolicited symptoms during the 31 days following vaccination and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 106345 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106345 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106345 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106345 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106345 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106345 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register